CLINICAL TRIAL: NCT06926842
Title: A Randomized, Double-Blind, Phase 2 Trial of Once-Weekly Petrelintide Compared With Placebo in Participants With Overweight or Obesity and Type 2 Diabetes
Brief Title: Efficacy and Safety of Petrelintide in Participants With Overweight or Obesity and Type 2 Diabetes (ZUPREME 2)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZP8396-24115
Record Dates: First submitted 2025-04-11; First posted 2025-04-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Type 2 Diabetes; Obesity
Keywords: Long-acting amylin analogues; Weight management
MeSH Terms: conditions — Overweight; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A: Petrelintide Dose 1 (Experimental): Randomized participants will receive weekly subcutaneous injections of petrelintide Dose 1.
  Interventions: Drug: Petrelintide
- Treatment B: Petrelintide Placebo Dose 1 (Placebo Comparator): Randomized participants will receive weekly subcutaneous injections of matching placebo to petrelintide.
  Interventions: Other: Placebo
- Treatment C: Petrelintide Dose 2 (Experimental): Randomized participants will receive weekly subcutaneous injections of petrelintide Dose 2.
  Interventions: Drug: Petrelintide
- Treatment D: Petrelintide Placebo Dose 2 (Placebo Comparator): Randomized participants will receive weekly subcutaneous injections of matching placebo to petrelintide.
  Interventions: Other: Placebo
- Treatment E: Petrelintide Dose 3 (Experimental): Randomized participants will receive weekly subcutaneous injections of petrelintide Dose 3.
  Interventions: Drug: Petrelintide
- Treatment F: Petrelintide Placebo Dose 3 (Placebo Comparator): Randomized participants will receive weekly subcutaneous injections of matching placebo to petrelintide.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Petrelintide — Petrelintide will be taken by participants once weekly subcutaneously.
  Other Names: ZP8396
  Arms: Treatment A: Petrelintide Dose 1; Treatment C: Petrelintide Dose 2; Treatment E: Petrelintide Dose 3
Other: Placebo — Matching placebo to petrelintide will be taken by participants once weekly subcutaneously.
  Arms: Treatment B: Petrelintide Placebo Dose 1; Treatment D: Petrelintide Placebo Dose 2; Treatment F: Petrelintide Placebo Dose 3

SUMMARY:
The main purpose of this study is to investigate efficacy and safety of three doses of petrelintide versus placebo in participants with overweight or obesity and type 2 diabetes.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female participants with body mass index (BMI) ≥27.0 kg/m2.
* Diagnosed with type 2 diabetes ≥180 days prior to the day of screening.
* Treated with metformin with or without sodium-glucose cotransporter 2 inhibitors. Treatment should be stable (same drug[s], dose, and dosing frequency) for at least 90 days prior to screening.

Main Exclusion Criteria:

* Severe hypoglycemia within 6 months prior to screening or history of hypoglycemia unawareness.
* Receipt of any other glucose-lowering drug than those listed in the inclusion criterion within 90 days prior to screening.
* A self-reported change in body weight >5% within 90 days prior to screening, irrespective of medical records.
* Treatment with any medication (prescribed or over-the-counter) or alternative remedies (herbal or nutritional supplements) intended to promote weight loss within 90 days prior to screening.
* Previous or planned (during the trial period) obesity treatment with surgery or a body weight loss device. However, liposuction or surgical removal of fat depots more than 1 year prior to screening or device-based interventions (e.g., sleeve, banding, or similar) that have been removed more than 6 months prior to screening, are allowed.
* Obesity due to endocrine disorders or genetic syndromes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-08-13 (Estimated); Study Completion 2026-08-13 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Body Weight | From Baseline (Day 1) to Weeks 28

SECONDARY OUTCOMES:
Number of Participants Achieving ≥5% Body Weight Loss | From Baseline (Day 1) to Weeks 28
Number of Participants Achieving ≥10% Body Weight Loss | From Baseline (Day 1) to Weeks 28
Change in Body Weight (kilogram) | From Baseline (Day 1) to Weeks 28
Change in Waist Circumference | From Baseline (Day 1) to Weeks 28
Change in Glycated Hemoglobin (HbA1c) | From Baseline (Day 1) to Weeks 28
Change in Fasting Glucose | From Baseline (Day 1) to Weeks 28
Change in High-Sensitivity C-reactive protein (hsCRP) | From Baseline (Day 1) to Weeks 28
Number of Participants Achieving ≤6.5% HbA1c | From Baseline (Day 1) to Weeks 28
Changes in Fasting Lipids | From Baseline (Day 1) to Weeks 28
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | From Baseline (Day 1) to Weeks 38
Number of Participants with Treatment- Emergent Severe or Clinically Significant Hypoglycemic Episodes from Baseline to Week 38 | From Baseline (Day 1) to Weeks 38
Number of Participants with Positive Anti-Drug Antibodies (ADAs) | From Baseline (Day 1) to Weeks 38
Change in Systolic Blood Pressure | From Baseline (Day 1) to Week 38
Change in Diastolic Blood Pressure | From Baseline (Day 1) to Week 38
Change in Pulse Rate | From Baseline (Day 1) to Week 38

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - Cullman Clinical Trials - Family Medicine, Cullman, Alabama
  - AZ Endocrine Institute, Chandler, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - M3 Wake Research, Tucson Neuroscience Research, LLC, Tucson, Arizona
  - Medical Investigation Inc, Little Rock, Arkansas
  - Velocity Clinical Research, Huntington Park, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Exalt Clinical Research, San Diego, California
  - Diablo Clinical Research Inc., Walnut Creek, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Emerson Clinical Research, Washington D.C., District of Columbia
  - Innovative Research of West Florida, Clearwater, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Solutions Through Advanced Research, Inc, Jacksonville, Florida
  - M3 Wake Research - Lake City, Lake City, Florida
  - West Orange Endocrinology P.A, Ocoee, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - M3 Wake Research - Atlanta, Atlanta, Georgia
  - East Coast Institute for Research - Canton, Canton, Georgia
  - Privia Medical Group Georgia, LLC, Savannah, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Iowa Diabetes & Endocrinology Research Center, West Des Moines, Iowa
  - Heartland Research Associates, LLC, Wichita, Kansas
  - DelRicht Research - New Orleans, New Orleans, Louisiana
  - AAMRC, Flint, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - Velocity Clinical Research, Gulfport, Gulfport, Mississippi
  - AMR Kansas City, Kansas City, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - M3 Wake Research - Las Vegas, NV, Las Vegas, Nevada
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Javara Inc, Charlotte, North Carolina
  - PharmQuest Life Sciences, LLC, Greensboro, North Carolina
  - M3 Wake Research, Raleigh, North Carolina
  - Velocity Clinical Research, Cincinnati, Mt. Auburn, Cincinnati, Ohio
  - Centricity Research, Columbus, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - M3 Wake Research - Charleston, Charleston, South Carolina
  - M3 Wake Research/ClinSearch, LLC, Chattanooga, Tennessee
  - Elligo Clinical Research, Inc., Austin, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Juno Research LLC, Houston, Texas
  - Tekton Research, LLC, Irving, Texas
  - Tekton Research, LLC, McKinney, Texas
  - Texas Health Care, PLLC, San Marcos, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Texas Health Care, Stephenville, Texas
  - Manaasas Clinical Research Center, Manassas, Virginia

IPD SHARING:
Plan to Share IPD: Undecided